CLINICAL TRIAL: NCT01155310
Title: An International Phase III Randomised Trial Comparing in Severe Exacerbations of Chronic Obstructive Pulmonary Disease the Efficacy of Helium/Oxygen Versus Air/Oxygen Administered During Spontaneous Breathing and Intermittent Non-Invasive Ventilation.
Brief Title: Efficacy of Helium/Oxygen Compared to Air/Oxygen in Severe Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)
Acronym: ECHO/ICU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: the observed event rate is lower than expected by the protocol hypothesis.
Sponsor: Air Liquide Santé International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALMED-07-C3-009
Record Dates: First submitted 2010-06-25; First posted 2010-07-01 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Exacerbation of COPD; Helium/Oxygen; ICU; Non-Invasive Ventilation; Patient with known or suspected COPD; patient Admitted in an ICU; Patient presenting current exacerbation of COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Helium; Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Helium/Oxygen (Experimental): Helium/Oxygen 78%/22% will be administered for a maximum of 72 hours.
  Interventions: Drug: Helium/Oxygen 78%/22%
- Air/Oxygen (Active Comparator): Air/Oxygen will be administered for a maximum of 72 hours.
  Interventions: Drug: Air/Oxygen

INTERVENTIONS:
Drug: Helium/Oxygen 78%/22% — The Helium/Oxygen mixture will be administered during NIV and NIV-free sessions for a maximum of 72 hours using study dedicated devices.
  Patients will then receive the Air/Oxygen mixture with usual devices.
  Arms: Helium/Oxygen
Drug: Air/Oxygen — The Helium/Oxygen mixture will be administered during NIV and NIV-free sessions for a maximum of 72 hours using study dedicated devices.
  Patients will then receive the Air/Oxygen mixture with usual devices.
  Arms: Air/Oxygen

SUMMARY:
The primary objective of the study is to evaluate the efficacy of Helium/Oxygen (He/O2) 78%/22% compared to a conventional Air/O2 mixture in reducing endotracheal intubation rate and mortality in patients with severe hypercapnic exacerbations of Chronic Obstructive Pulmonary Disease (COPD) during their index Intensive/Intermediate Care Unit (ICU) stay.

DETAILED DESCRIPTION:
Patients eligible for this study are critically ill patients with COPD admitted in Intensive Care Unit for an exacerbation of their chronic disease with hypercapnic acute respiratory failure. The patients will receive an Helium/Oxygen mixture or an Air/Oxygen mixture for a maximum of 72 hours during Non-Invasive Ventilation (NIV) and NIV-free sessions.

During NIV sessions, gas mixtures will be administered using a ventilator suitable for NIV with either He/O2 or Air/O2 and a NIV facemask.

Patients will be followed until hospital discharge and then contacted by phone up to the 6th month after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient with known or suspected COPD
* Patient presenting current exacerbation of COPD with hypercapnic acute respiratory failure
* Patient eligible for Non-Invasive Ventilation (NIV)
* Patient admitted in an ICU

Exclusion Criteria:

* Patient who had lung transplant
* Patient having a contraindication to NIV
* Patient with tracheostomy
* Patient requiring Oxygen flow rate > 6 L/min or Inspired Oxygen Fraction (FIO2) > 0.50
* Patient admitted in the ICU for more than 24 hours and/or having received NIV in ICU for more than 6 hours (in total) for the current exacerbation of COPD

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2010-05; Primary Completion 2013-10 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Reduction of NIV failure | 10 days (average)
  Endotracheal intubation and/or death

SECONDARY OUTCOMES:
Duration of ICU stay and duration of index hospitalisation | 10 days (average)
Duration of invasive ventilation | 10 days (average)
Adverse events | 6 months (post-randomization)
Medico-economic parameters | 6 months
  Overall costs and cost-effectiveness
Physiological and laboratory parameters | 10 days (average)
  Systolic and diastolic blood pressures, heart rate, central body temperature, arterial oxygen saturation, haematology and serum biochemistry
Duration of NIV sessions | 10 days (average)
  Cumulative daily duration of NIV sessions and their number during each of the 3-day treatment period and globally
Time interval between the discharge of the index ICU stay and the first re-admission in ICU for severe exacerbation of COPD | 6 months (post-randomization)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe JOLLIET, Prof., Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (16):
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - Les Cliniques Universitaires UCL Mont Godinne, Yvoir
- France (9):
  - Centre Hospitalier Universitaire Angers, Angers
  - Centre Hospitalier Universitaire Pellegrin-Tripode, Bordeaux
  - Hôpitaux de Chartes, Chartres
  - CHU Clermont-Ferrand - Hôpital ESTAING, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CHU NICE - Hopital Pasteur, Nice
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer - Hopital Sainte Musse, Toulon
- Azienda Ospedaliera Univeritaria Careggi, Florence, Italy
- Hôpitaux Universitaires de Genève, Geneva, Switzerland
- Tunisia (2):
  - Hôpital Abderrahmen Mami, Aryanah
  - Centre Hospitalier Universitaire Fattouma Bourguiba, Monastir
- University Hospital of North Tees, Stockton-on-Tees, United Kingdom

REFERENCES:
- [Derived] Jolliet P, Ouanes-Besbes L, Abroug F, Ben Khelil J, Besbes M, Garnero A, Arnal JM, Daviaud F, Chiche JD, Lortat-Jacob B, Diehl JL, Lerolle N, Mercat A, Razazi K, Brun-Buisson C, Durand-Zaleski I, Texereau J, Brochard L; E.C.H.O. ICU Trial Investigators. A Multicenter Randomized Trial Assessing the Efficacy of Helium/Oxygen in Severe Exacerbations of Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2017 Apr 1;195(7):871-880. doi: 10.1164/rccm.201601-0083OC. PMID 27736154